CLINICAL TRIAL: NCT05415956
Title: "Outwalk MS" - Benefits of Outdoor Walking Exercise Therapy on Walking Capacity and Well-being in Multiple Sclerosis
Brief Title: "Outwalk MS" - Benefits of Outdoor Walking in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish MS Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Outwalk_MS
Record Dates: First submitted 2021-11-25; First posted 2022-06-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2021-11

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Walking
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 7 week randomized controlled trial; intervention group and waitlist/control group.
  The investigators will perform a cluster randomization (computer generated random numbers) according to cities across Denmark (when 4-12 pwMS are interested and eligible).
  Waitlist/control group will be offered the same outdoor walking exercise therapy after the initial 7 weeks.
  24 weeks after the walking exercise intervention, a follow-up test will be carried out as well.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking exercise therapy (Experimental): 7 week intervention group. 6-12 persons per group. 2 sessions per week, 14 sessions in total.
  Surface: the investigators aim to involve as much forest/gravel trails as possible, with up/down hill walking.
  Uneven session numbers: warm-up (6 minutes at BORG 10-11), continous walking (starting at 12-20 minutes at BORG 13-14 and progressing to 20-40 minutes at BORG 15-16, adjusted according to the starting level of each participant) and cool-down (approximately 10 minutes at BORG 10-11).
  Even session numbers: warm-up (6 minutes at BORG 10-11), intermittent walking (starting at 3-4 intervals of 2 minutes at BORG 14-15 and progressing to 4-5 intervals of 2-3 minutes at BORG 16-17; with all intervals being interspersed by 1 minute rest) and cool-down (approximately 10 minutes at BORG 10-11).
  Interventions: Behavioral: Walking exercise therapy
- Control/Waitlist (No Intervention): 7 week control/waitlist group. Continuation of habitual lifestyle during the 7 week intervention period (yet these participants will receive the exact walking exercise therapy afterwards).

INTERVENTIONS:
Behavioral: Walking exercise therapy — Moderate-to-high intensity walking exercise therapy (7 weeks, 14 session) with progression in duration and intensity.
  Other Names: Physical exercise
  Arms: Walking exercise therapy

SUMMARY:
Deterioration of walking capacity is a common symptom in persons with multiple sclerosis (pwMS), furthermore having a negative influence on well-being. Studies have nevertheless shown that walking exercise therapy can improve walking capacity in pwMS. This may be particularly potent if occurring outdoors due to the varying stimuli it can provide (different surfaces and terrain etc.), and if the intensity and duration is adequate. Furthermore, outdoor walking is (1) suitable as a group intervention facilitating interaction between pwMS and (2) advantageous due to the health benefits offered through the interaction with nature itself. Both these aspects are also relevant for well-being.

Few studies have nevertheless examined the effects of outdoor walking exercise therapy in pwMS. The purpose of the present study is therefore to examine the effects of 7 weeks of moderate-to-high intensity outdoor walking exercise therapy on walking capacity (primary outcome: 6-minute walk test) and well-being in pwMS.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* self-reported clinical MS diagnosis
* PDDS ≤ 4 (corresponding to preserved walking capacity without assistive devices of at least 10 m)
* able to independently attend the testing

Exclusion Criteria:

* self-reported comorbidities excluding participation in the intervention
* recent (6 months retrospective) fractures, amputation or other critical physical impairments that eliminates participation in the described training study
* participation in structured exercise therapy (including walking) for the past 3 months (≥ 2 session per week of moderate-to-high intensity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
6-minutes walk test (6MWT) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Maximal distance covered in 6 minutes using a 30 meter walkway. Assesses walking endurance.

SECONDARY OUTCOMES:
6-minutes walk test (6MWT) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Maximal distance covered in 6 minutes using a 30 meter walkway. Assesses walking endurance.
Timed 25-foot walk test (T25FWT) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Time used to complete a 25-foot (= 7.62 meters) walk test. Two trials are given. Assesses horizontal walking propulsion/acceleration (i.e. walking speed).
Timed 25-foot walk test (T25FWT) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Time used to complete a 25-foot (= 7.62 meters) walk test. Two trials are given. Assesses horizontal walking propulsion/acceleration (i.e. walking speed).
Six spot step test (SSST) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Time used to complete the SSST (5 wooden blocks must be pushed/kicked outside their initial position). Four trials are given, two with each foot being used to push/kick the wooden blocks. Assesses horizontal coordination and dynamic balance during walking.
Six spot step test (SSST) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Time used to complete the SSST (5 wooden blocks must be pushed/kicked outside their initial position). Four trials are given, two with each foot being used to push/kick the wooden blocks. Assesses horizontal coordination and dynamic balance during walking.
12-item multiple sclerosis walking scale (MSWS-12) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing patient-reported impact of multiple sclerosis on walking ability.
  Total score range 12-60 (0-100%); lower is better.
12-item multiple sclerosis walking scale (MSWS-12) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing patient-reported impact of multiple sclerosis on walking ability. 12 questions.
  Total score range 12-60 (0-100%); lower is better.
Modified fatigue impact scale (MFIS) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing patient-reported perceived fatigue impact. 21 questions.
  Total score range 0-84; lower is better. Physical subscale score range (9 questions) 0-36; lower is better. Cognitive subscale score range (10 questions) 0-40; lower is better. Psychosocial subscale score range (2 questions) 0-8; lower is better.
Modified fatigue impact scale (MFIS) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing patient-reported perceived fatigue impact. 21 questions.
  Total score range 0-84; lower is better. Physical subscale score range (9 questions) 0-36; lower is better. Cognitive subscale score range (10 questions) 0-40; lower is better. Psychosocial subscale score range (2 questions) 0-8; lower is better.
Falls-efficacy scale (FES-I) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing concerns of falling along with history of falls.
  7 questions. Total score range 0-28; lower is better. History of falls: one year recall.
Falls-efficacy scale (FES-I) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing concerns of falling along with history of falls.
  7 questions. Total score range 0-28; lower is better. History of falls: one year recall.
WHO five well-being index (WHO5) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing patient-reported well-being. 5 questions. Score range 0-25 (0-100%); higher is better.
WHO five well-being index (WHO5) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing patient-reported well-being. 5 questions. Score range 0-25 (0-100%); higher is better.
EuroQoL 5 dimensions 3 levels (EQ5D) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing patient-reported quality of life.
  VAS scale score range 0-100%; higher is better. 5 domains, scored separately, score range 1-3; lower is better.
EuroQoL 5 dimensions 3 levels (EQ5D) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing patient-reported quality of life.
  VAS scale score range 0-100%; higher is better. 5 domains, scored separately, score range 1-3; lower is better.
Baecke physical activity questionnaire | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing patient-reported participation in physical activities.
  4 questions. Score range is continuous (0-xx). Higher is better.
Baecke physical activity questionnaire | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing patient-reported participation in physical activities.
  4 questions. Score range is continuous (0-xx). Higher is better.
Patient-determined disease steps (PDDS) | Change from baseline (Pre) to after 7 weeks intervention (Post)
  Questionnaire (patient-reported outcome) assessing patient-reported disability in multiple sclerosis (MS).
  9 questions/categories. Each category represents disability level; lower is better.
Patient-determined disease steps (PDDS) | Change from baseline (Pre) to 24 weeks follow-up (Follow-up)
  Questionnaire (patient-reported outcome) assessing patient-reported disability in multiple sclerosis (MS).
  9 questions/categories. Each category represents disability level; lower is better.

CONTACTS AND LOCATIONS:
Overall Officials: Lars G Hvid, MSc, PhD, Principal Investigator — Aarhus University, Department of Public Health, Exercise Biology
Locations (1):
- Aarhus University, Health, Exercise Biology, Aarhus, Jutland, Denmark

REFERENCES:
- [Derived] Hvid LG, Steenberg JL, Roy F, Skovgaard L. Outdoor walking exercise therapy improves walking capacity and well-being in persons with multiple sclerosis: A randomized controlled trial. Ann Phys Rehabil Med. 2025 Sep;68(6):101985. doi: 10.1016/j.rehab.2025.101985. Epub 2025 Apr 18. PMID 40252300